CLINICAL TRIAL: NCT06525623
Title: Initial Resuscitation for Acute Kidney Injury in Patients With Cirrhosis: A Pilot Randomized Trial Using a Volume Assessment Guidance Algorithm
Brief Title: Initial Resuscitation for Acute Kidney Injury in Cirrhosis
Acronym: RAKI-VAGA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Andrew S. Allegretti, MD, MSC, Director of Critical Care Nephrology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024P001520; K23DK128567 (NIH)
Record Dates: First submitted 2024-07-16; First posted 2024-07-29 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Cirrhosis, Liver; Acute Kidney Injury; Hepatorenal Syndrome
MeSH Terms: conditions — Liver Cirrhosis; Acute Kidney Injury; Hepatorenal Syndrome | interventions — Crystalloid Solutions; Colloids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VAGA Group (Experimental): This group will receive an algorithm-based recommendation based on the 2024 Acute Disease Quality Initiative (ADQI)/International Club of Ascites (ICA) joint consensus meeting on AKI in cirrhosis, which recommends a personalized approach to AKI in cirrhosis in order to avoid volume overload. This includes balanced crystalloids as first-line resuscitative fluids unless there is a patient-specific indication for an alternative colloid (e.g. blood for gastrointestinal bleeding, IV albumin for spontaneous bacterial peritonitis or suspicion of hepatorenal syndrome), or no further resuscitation.
  Interventions: Other: Recommendation: No Further Resuscitation; Other: Recommendation: Resuscitation with Crystalloid; Other: Recommendation: Resuscitation with Colloid
- Standard of Care (Placebo Comparator): This group will receive a recommendation based on the 2021 American Association for the Study of Liver Diseases (AASLD) and 2018 European Association for the Study of the Liver (EASL) clinical practice guidelines, which recommends a 1 g/kg/d IV albumin (maximum 100 g/day) IV albumin over 2 days as an initial resuscitation approach for patients with AKI and cirrhosis.
  Interventions: Other: Recommendation: Standard of Care IV Albumin

INTERVENTIONS:
Other: Recommendation: No Further Resuscitation — Treatment teams are encouraged not to administer any additional fluids
  Arms: VAGA Group
Other: Recommendation: Resuscitation with Crystalloid — Treatment teams are encouraged to administer crystalloid. Amount of resuscitative fluid will be determined by treatment team's clinical assessments and usual standards of care
  Arms: VAGA Group
Other: Recommendation: Resuscitation with Colloid — Treatment teams are encouraged to administer colloid. Amount of resuscitative fluid will be determined by treatment team's clinical assessments and usual standards of care
  Arms: VAGA Group
Other: Recommendation: Standard of Care IV Albumin — Treatment teams are encouraged to administer 1 g/kg/d IV albumin (maximum 100 g/day) over 2 days
  Arms: Standard of Care

SUMMARY:
The goal of this interventional study is to evaluate two strategies for how to provide intravenous (IV) fluids for treating patients with acute kidney injury (AKI) in cirrhosis. The main question it aims to answer is: what is the safety, efficacy, and feasibility of providing a recommendation to use a Volume Assessment Guidance Algorithm (VAGA) or give standard of care doses of IV albumin?

Patients will be randomly assigned where their treating teams will receive a VAGA-based recommendation or a standard of care IV albumin recommendation.

DETAILED DESCRIPTION:
This randomized, open-label, pilot feasibility trial will assess a volume assessment guidance algorithm (VAGA) in patients with AKI and cirrhosis. Eligible patients must have AKI and decompensated cirrhosis. In addition to assessing the adherence to the suggested guidance, this study will measure the effect of the study intervention on grams of albumin given, clinical efficacy outcomes (AKI response rates, survival, RRT status, transplant status), and safety.

Patients who meet eligibility criteria will be randomized 1:1 where the treating clinicians will receive a one-time recommendation for volume resuscitation using the VAGA or standard of care IV albumin repletion (1 g/kg/day for two days). Both groups will be followed with assessments at 48 hours after randomization, hospital discharge, and 90-days after randomization.

The primary efficacy outcome, grams of albumin, will be measured at 48 hours after randomization. Primary secondary efficacy outcomes (grams of albumin, AKI response) will be assessed at time of hospital discharge. If a patient undergoes liver transplantation or initiation of RRT during the admission, this will serve as a censoring date for these outcomes, and relevant data will be collected at the time of the first of these events.

The primary feasibility outcome is adherence to the suggested guidance, assessed at 48 hours after randomization. The VAGA group will receive one of three potential clinical recommendations: (a) no further volume resuscitation, (b) resuscitation with crystalloid, or (c) resuscitation with colloid.

This study will prospectively enroll approximately 50 adult patients at a single center.

ELIGIBILITY:
Inclusion Criteria:

1. Adult age 18 years or greater
2. Signed informed consent form (ICF) by any subject capable of giving consent, or, when the subject is not capable of giving consent, by their legally authorized representatives prior to initiation of any study procedures.
3. Admitted to the hospital
4. Diagnosis of decompensated cirrhosis (either prior to admission or new diagnosis on admission).
5. Presence of acute kidney injury (AKI) as defined by International Club of Ascites (ICA) criteria, defined as SCr increase of ≥0.3 mg/dL within 48 hours or ≥50% increase from baseline which is known or presumed to have occurred within the prior 7 days.

Exclusion Criteria:

1. Requiring >2 liters (L) supplemental oxygen at the time of screening.
2. In shock requiring vasopressors (vasoconstrictors for the treatment of AKI such as terlipressin, midodrine, and octreotide are allowed).
3. Allergy or other contraindication to IV albumin administration.
4. Death, liver transplant, or renal replacement therapy (RRT) expected within 48 hours.
5. Patient and/or legally authorized representative unable to provide informed consent.
6. Hepatic encephalopathy grade 3 or 4 at the time of screening.
7. Already received >200 g albumin during admission at the time of screening.
8. Severe, active bleeding requiring 3 or more units of red blood cell transfusion in the 48 hours prior to screening.
9. Admission to the intensive care unit at the time of screening.
10. Mechanical ventilation at the time of screening.
11. Presence of New York Heart Association (NYHA) class 3-4 symptoms of congestive heart failure at the time of screening.
12. History of prior liver or kidney transplant.
13. Pregnant or nursing status
14. Any condition, in the opinion of the investigator, that could confound or interfere with the safe completion of study activities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
IV albumin received (grams) | From date of randomization up to 48 hours
Adherence to suggested guidance | From date of randomization up to 48 hours
  For the VAGA group, adherence is defined as: No further resuscitation (<500 mL total volume of IV fluid given), Resuscitation with crystalloid (>500 mL total IV fluid given, with <50 g IV albumin and ≤2 units blood), Resuscitation with colloid (≥50 g IV albumin or ≥2 units blood given). For the Standard of Care group, adherence is defined as receiving within 20% of the suggested IV albumin dose in grams.
Incidence of treatment-emergent adverse events and serious adverse events | From date of randomization up to hospital discharge, assessed up to 90 days

SECONDARY OUTCOMES:
IV albumin received (grams) | From date of hospital admission up to hospital discharge, or the date of time of initiation of renal replacement therapy or liver transplant, whichever came first, assessed up to 90 days.
AKI Response | From date of randomization up to hospital discharge, or the date of time of initiation of renal replacement therapy or liver transplant, whichever came first, assessed up to 90 days.
  AKI response is defined as complete response (return of serum creatinine to a value within 0.3 mg/dL of the baseline value), partial response (regression of AKI stage with a reduction of serum creatinine (SCr) to ≥0.3 mg/dl above the baseline value), or no response (neither complete or partial response met).
Vital Status | From date of randomization up to 90 days
  Alive or dead
Renal Replacement Therapy Initiation | From date of randomization up to 90 days
  Yes or No
Liver transplant | From date of randomization up to 90 days
  Yes or No

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Intellectual property and data generated under this project will be administered in accordance with both Massachusetts General Hospital and NIH policies, including the NIH Data Sharing Policy and Implementation Guidance of March 5, 2003.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After the final research data set has been accepted for publication for 1 year.
Access Criteria: Upon request

REFERENCES:
- [Background] European Association for the Study of the Liver. EASL Clinical Practice Guidelines for the management of patients with decompensated cirrhosis. J Hepatol. 2018 Aug;69(2):406-460. doi: 10.1016/j.jhep.2018.03.024. Epub 2018 Apr 10. No abstract available. PMID 29653741
- [Background] Biggins SW, Angeli P, Garcia-Tsao G, Gines P, Ling SC, Nadim MK, Wong F, Kim WR. Diagnosis, Evaluation, and Management of Ascites, Spontaneous Bacterial Peritonitis and Hepatorenal Syndrome: 2021 Practice Guidance by the American Association for the Study of Liver Diseases. Hepatology. 2021 Aug;74(2):1014-1048. doi: 10.1002/hep.31884. No abstract available. PMID 33942342
- [Background] Nadim MK, Kellum JA, Forni L, Francoz C, Asrani SK, Ostermann M, Allegretti AS, Neyra JA, Olson JC, Piano S, VanWagner LB, Verna EC, Akcan-Arikan A, Angeli P, Belcher JM, Biggins SW, Deep A, Garcia-Tsao G, Genyk YS, Gines P, Kamath PS, Kane-Gill SL, Kaushik M, Lumlertgul N, Macedo E, Maiwall R, Marciano S, Pichler RH, Ronco C, Tandon P, Velez JQ, Mehta RL, Durand F. Acute kidney injury in patients with cirrhosis: Acute Disease Quality Initiative (ADQI) and International Club of Ascites (ICA) joint multidisciplinary consensus meeting. J Hepatol. 2024 Jul;81(1):163-183. doi: 10.1016/j.jhep.2024.03.031. Epub 2024 Mar 26. PMID 38527522